CLINICAL TRIAL: NCT06526689
Title: Investigating the Impact of the Pulmonary Innate Immune Response and Microbiome After Exposure to Mycobacterium Tuberculosis
Brief Title: Lung Innate Immunity and Microbiome After Tuberculosis Exposure
Acronym: LIMBO-TB
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: LIMBO-TB
Record Dates: First submitted 2024-05-15; First posted 2024-07-30 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis; Latent Tuberculosis
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples Sputum Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Adult volunteers who are recent contacts of Mycobacterium tuberculosis sputum smear positive cases with positive IGRA
- Group B: Adult volunteers who are recent contacts of Mycobacterium tuberculosis sputum smear positive cases with negative IGRA
- Group C: Healthy adult volunteers with no previous exposure to Mycobacterium tuberculosis.

SUMMARY:
To characterise the innate pulmonary immune response and respiratory microbiome after recent exposure to M.tb and to evaluate how differences determine the outcome of M.tb exposure

DETAILED DESCRIPTION:
Tuberculosis (TB) kills more people than any other single infectious disease. It is estimated that 1 in 4 people are infected with the bug that causes TB. We really need an effective vaccine to prevent people getting TB, but we don't understand what sort of immune response is needed to protect people.

The very early response to infection, called the innate immune response, is not well understood in TB, partly because it is difficult to study, as most of the changes happen before people get symptoms. In a recent study we have seen that human infection with BCG, a bacteria similar to the one that causes TB, results in significant changes in the early immune response in the lungs, which are not seen in the blood.

The immune system is constantly coming into contact with different bacteria which live on the surfaces of our bodies, called the microbiome, this includes the linings of the airways (the tubes of the lungs). Understanding the interactions between the microbiome in the airways and immune system can help us to understand why some people can resist developing TB.

This study has been designed to help to answer two key questions about the early immune responses to TB:

1. What is the early immune response to TB, and how does it vary between people? We will use samples of sputum from people who have recently been living with someone with an active TB infection. We will measure the type of immune cells present in these samples and how they change over time, comparing what we find with blood results. This will help us to build a picture of what is happening both in the airways and in the blood during the early immune responses to TB.

   The immune response to TB is also different in different people. Importantly, some people never develop a memory (or 'adaptive') immune response. This may suggest that the early immune response is able to clear all of the infection quickly in these people. Understanding differences in the early immune response would give us ways to develop more effective vaccines and treatments.
2. Does the microbiome of the airway help in protecting people from TB? The bacteria of the microbiome live in unison with our cells, and are able to survive without causing an infection which makes us unwell. It has increasingly been understood that these bacteria help to "train" our immune system to work better. We will look at which bacteria are living normally in the airways of the people recruited to our study, and see how these bacteria change over time. This will help us to get a greater understanding of how the immune system and the microbiome work together, and if there is a role for the microbiome in preventing TB infections.

In summary this study will look at the early immune responses and the airway microbiome of people who have recently come into contact with the bacteria which causes TB. The differences that we identify could help us explain why some people have protection from TB, and provide us with novel approaches to developing new ways to protect others.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years
2. Resident in or near London or Oxford for the duration of the study period
3. Provide written informed consent
4. Willing to allow the investigators to review the volunteer's review NHS care record, medical history, blood results and radiographs.
5. Able and willing (in the investigator's opinion) to comply with all study requirements

   Group A and B Specific Inclusion Criteria
6. Have undergone screening for TB through NHS services (including IGRA testing +/- CXR where indicated)
7. Close contact with a sputum smear positive TB case within the last 12 weeks

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment or during the trial follow up period.
2. History of anaphylaxis or any allergy likely to be exacerbated by any essential study procedure
3. History of currently poorly controlled of airways disease (including asthma), current cancer (except BCC of the skin or CIS of the cervix), bleeding disorder, or drug or alcohol abuse
4. Any significant autoimmune conditions or immunodeficiency (including HIV)
5. Previous diagnosis or treatment for TB disease or latent TB infection
6. Clinical, radiological, or laboratory evidence of current active TB disease
7. Previous receipt of any investigational TB vaccines or aerosolised BCG.
8. Clinically Significant abnormalities in spirometry.
9. Concurrent use of oral, inhaled or systemic steroid medication or use for more than 14 days within the last 6 months (steroids used as a cream or ointment are permissible), or the use of other immunosuppressive agents concurrently or for more than 14 days within the last 6 months
10. Use of antibiotics in the past 4 weeks.
11. Administration of immunoglobulins and/or any blood products within the three months preceding the planned study
12. Administration of a live vaccine within the preceding 28 days prior to enrolment.
13. Administration of any other non-live vaccine within the preceding 14 days prior to enrolment.
14. Pregnancy or intention to become pregnant during study period
15. Any other significant disease, disorder, or finding, which, in the opinion of the investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the study or impair interpretation of the study data

    Group C Specific Exclusion Criteria
16. History of close contact with case of TB, or previous contact tracing by TB services.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human Adults with and with our recent exposure to M.tb
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The immunological response after recent M.tb exposure measured as the differentials of innate immune cells in the blood and sputum. | At enrolment and Day 84
  We will characterise the number and activity of early immunological response to M.tb in the respiratory tract and systemic circulation. Samples of blood and sputum will be utilised to enumerate the proportions of innate immune cells measured by flow cytometry and their activity.

SECONDARY OUTCOMES:
An assessment of respiratory microbiome diversity in M.tb contacts compared to healthy controls | At enrolment and Day 84
  To characterise the respiratory microbiome after exposure to M.tb by identifying bacterial genetic sequences and calculating both alpha diversity and beta diversity of sputum samples. Baseline and followup sample at day 84 will be investigated to determine robustness of communities.

OTHER OUTCOMES:
Exploratoring the role of innate immune response and microbiome on determining infection status by M.tb | At enrolment and Day 84
  We will combine data on the microbial communities identified in sputum as well as their diversity and combine it with data on the innate immune responses to explore whether measurements can be used to predict latent TB infection.
  Utilised assays may include but will not be limited to:
  Flow cytometry ELISAs Ellispots Sequencing data of bacterial isolates from sputum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, PhD, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Churchill Hospital, Oxford, Oxfordshire
  - Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxon
  - Grove Building, Royal Free NHS Foundation Trust, London

DOCUMENTS (1):
  • Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT06526689/ICF_000.pdf